CLINICAL TRIAL: NCT03898726
Title: Comparison Between Laparoscopic Versus Transvaginal Cuff Closure After Total Laparoscopic Hysterectomy
Brief Title: Laparoscopic Versus Transvaginal Cuff Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El-Galaa Military Medical Complex (Other Government)
Responsible Party: Principal Investigator, amr saad mahmoud, assistant lecturer, El-Galaa Military Medical Complex
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ElGalaa
Record Dates: First submitted 2019-03-21; First posted 2019-04-02 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Vaginal Cuff Dehiscence; Vaginal Hematoma; Vaginal Infection
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: neither the paticipant nor the investigator knew type of vaginal cuff closure
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopical l cuff closure (Active Comparator): needle holder laparoscopic vaginal cuff closure
  Interventions: Biological: laparoscopical l cuff closure
- transvaginal cuff closure (Active Comparator): transvaginal cuff closure
  Interventions: Biological: laparoscopical l cuff closure

INTERVENTIONS:
Biological: laparoscopical l cuff closure — closure of vaginal cuff following hysterectomy
  Other Names: transvaginal cuff closure

SUMMARY:
It is still debatable whether that the transvaginal approach to vault closure or laparoscopic suturing are associated with lower risks of vaginal cuff complications .

This study aims to compare the two approaches of closure of the vaginal cuff at the end of total laparoscopic hysterectomy as regards the vaginal cuff complications .

DETAILED DESCRIPTION:
All the women will subject to:

Preoperative Assessment including:

* Detailed history taking including age ,parity, medical ,surgical history .
* Physical examination:

  * General examination including the body mass index .
  * Abdominal examination including presence of previous scars, uterine size , any tenderness and presence of palpable masses .
  * Pelvic examination: including uterine size, any adnexal mass and tenderness .
* Preoperative investigation:

  * A preoperative trans-vaginal ultra- sonography to assess the volume of the uterus, gross uterine pathology and any adnexal pathology.
  * The preoperative laboratory investigation: hemoglobin percent and haematocrit value, blood grouping ,liver and kidney function tests.

Availability of blood was ensured for each patient before surgery.

Anaesthesia:

Standardized general anaesthetic technique consisting of induction agent, muscle-relaxant and inhalational agents with basic minimum monitoring after a detailed pre-anaesthetic check-up and adequate premedication advice.

Intraoperative :

* For vaginal cuff closure both in laparoscopic approach and vaginal route, the investigators will use the horizontal method, which can be described as closing the vagina anterior to posterior by leaving a horizontal scar. The repair will start at one end of the vaginal cuff, and will continue toward the surgeon , using a continuous Vicryl suture .
* In the laparoscopic approach, needles will be introduced through one trocar and removed through the opposite trocars using a needle holders.

Postoperative care:

1. The patient will receive IV fluids in the first 24hours (3litres).
2. Oral clear fluid intake will be started 8 hours after the operation.
3. Another dose of antibiotics will be received 6hrs after the operation with the same regimen used in induction.
4. Postoperative analgesia will be received in the form of parental NSAIDs every 8hrs for 24hrs then on demand.
5. The urinary catheter and the vaginal pack will be removed 24hrs after the operation , no drains will be left intraoperative.
6. CBC will be done 24hrs after the operation.
7. Histopathological examination of the specimen will be done.
8. Precocious resumption of coital activity ,( all patients will be recommended to avoid vaginal intercourse for at least 2 months ) .

Follow Up:

* Transvaginal ultrasound will be done to all patients in the second day to Spot vaginal cuff hematoma if found .
* Women will be discharged on antibiotic ( third generation cephalosporins ) and analgesics ( NSAIDs ) and a follow-up visit will be scheduled after 7 days for a full examination to exclude vaginal cuff infection ( purulent drainage from the vaginal cuff on gross anatomic exam according to CDC ) or cuff hematoma (Any blood collection at the level of vaginal vault detected by transvaginal ultrasound).
* All women will be followed up after 3 months for the occurrence of vaginal cuff dehiscence (separation of a vaginal incision that was previously closed at time of initial hysterectomy) , at that time all women will undergo abdominal examination and bimanual pelvic examination for vaginal masses.
* All women will be asked for dyspareunia according to Marinoff scale:

  0= no pain with intercourse .
  1. pain with intercourse that doesn't prevent the completion .
  2. pain with intercourse requiring interruption or discontinuance .
  3. pain with intercourse preventing any intercourse .
* Ethical Considerations:
* Patient information and informed consent:

Before being admitted to the clinical study, the patient must consent to participate after the nature, scope and possible consequences of the clinical study have been explained in a form understandable to her.

Protocol approval:

Before the beginning of the study and in accordance with the local regulation followed, the protocol and all the corresponding documents will be declared for Ethical and Research approval by the council of the OB/GYN department, Ain Shams University.

Assessment of the outcomes:

Primary outcomes:

1. Vaginal cuff dehiscence: Any separation at the level of the vaginal vault.

Secondary outcomes:

1. Vaginal cuff hematoma:

   Any blood collection at the level of vaginal vault detected by transvaginal ultrasound.
2. Post operative pelvic infections:

   Any postoperative infection with signs and symptoms of vaginal cuff involvement including granulation formation .
3. Operative time:

   Time spent in suturing the vaginal cuff transvaginally versus laparoscopically .
4. Incidence of dyspareunia : according to Marinoff scale .

ELIGIBILITY:
Inclusion Criteria:

1. Patients candidate for total laparoscopic hysterectomy :

   * Uterine size <12 weeks.
   * Having no severe endometriosis.
   * Having descent of no more than 1st degree of uterus.
   * Non-malignant conditions.
2. Completion of the entire procedure by laparoscopic approach up to colpotomy.
3. Benign conditions as indications for hysterectomy.

Exclusion Criteria:

- 1) Obese patients i.e., BMI > 30 k.g\m2. 2) Suspected extensive pelvic adhesions . 3) Factors which may prolong wound healing as uncontrolled diabetes, ,prolonged corticosteroid therapy ,advanced liver diseases.

4) Inability to express adequate informed consent to participate in the study.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
1. number of cases ofVaginal cuff dehiscence | 3 months
  Any separation at the level of the vaginal vault.

SECONDARY OUTCOMES:
number of cases with vaginal hematoma | 3 months
  ultrasound finding
number of cases with vaginal infection | 3 months
  purulent vaginal discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided